CLINICAL TRIAL: NCT02339480
Title: Research on Mechanism of Massage Therapy on Energy Metabolism Disorder of Simple Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guiyang College of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20141021
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Simple Obesity
Keywords: Massage therapy; Simple obesity; Energy metabolism; Mechanism
MeSH Terms: interventions — Massage

ARMS (2):
- Healthy volunteers (No Intervention): Healthy volunteers'hypothalamus picture of fMRI will compare with Obesity group' , no intervention and remaining unchanged lifestyle.
- Obesity group (Active Comparator): An intervention group of patients is put on a waiting list for massage therapy.Observing the Curative effect and hypothalamus picture of fMRI compare with healthy volunteers
  Interventions: Other: Massage therapy

INTERVENTIONS:
Other: Massage therapy — Healthy volunteers do not accept treatment, just to be a control group to compare with obesity group
  Arms: Obesity group

SUMMARY:
This project is to penetrate and consummate the research mechanism of massage therapy on simple obesity. Latest researches indicate that the energy regulation network system of hypothalamus and metabolic disorders on adipocyte may be the pathological bases which result in obesity. The research group have firstly conducted effect studies of massage therapy on model of simple obesity rats and observed some neurobiological mechanism (whole effect mechanism), meanwhile, the team have discussed influences on the development of preadipocyte and function of endocrine with dynamic mechanical stimulation in vitro (local effect mechanism). This research aims at centering on the hypothesis that massage therapy can act on energy regulation network system of hypothalamus specifically, thus regulating the energy metabolic disorders. Then applying functional magnetic resonance imaging (fMRI) to explore whether patients with simple obesity exist abnormality on energy regulation network system of hypothalamus, ascertain mechanisms how massage therapy treat energy metabolism disorders of simple obesity, deepen mechanism study on how massage therapy prevent and treat obesity and enrich the clinical application's scientific connotation that massage therapy treat simple obesity.

DETAILED DESCRIPTION:
This project will divide in two groups,healthy volunteers and obesity group.Healthy volunteers do not accept any treatment while obesity group need accept massage therapy three times a week,18 times in total.And two groups will be checked by functional magnetic resonance imaging (fMRI), Healthy volunteers for once and obesity group for twice(before treatment, obesity group's image of fMRI will compare with Healthy volunteers' and the image which is taken after treatment)

ELIGIBILITY:
Inclusion Criteria:

1.above 20% of the normal weight;BMI≥25.0；F%≥30%;

2.18-60 years old；

3.Patients agreeing and signing the Informed Consent for the study．

Exclusion Criteria:

1. The individuals do not adhere to the treatment or are with other treatments.
2. Secondary obesity, eg:pituitary diseases, hypothalamic disorder, hypothyroidism, pancreatic diseases，hyperadrenocorticism, postmenopausal obesity etc.
3. Having therapy for obesity in the last two weeks.
4. The individuals with server cardiovascular and cerebrovascular diseases and cancer.
5. Critical patients or patients combined with liver and kidney damage.
6. Individuals with psychosis.
7. Female individuals with pregnancy, lactation and planning a pregnancy in the two months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
body mass index(BMI) | 6 weeks after treatment

SECONDARY OUTCOMES:
Body Weight | 6 weeks after treatment
waistline | 6 weeks after treatment
hip line | 6 weeks after treatment
thigh line | 6 weeks after treatment
percentage of body fat | 6 weeks after treatment

OTHER OUTCOMES:
image of hypothalamus of functional magnetic resonance imaging (fMRI) | before treatment and 6 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Guiyang College of Troditional Chinese Medicine, Guiyang, Guizhou, China